CLINICAL TRIAL: NCT01597167
Title: A Double-blinded Randomized Study of IV Infusion of Magnesium Sulfate Versus 5% Dextrose in a Crossover Design in Male and Female Volunteers With Treatment Resistant Depression
Brief Title: Magnesium Sulfate Versus 5% Dextrose With Treatment Resistant Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Life Extension Foundation Inc. (Other)
Responsible Party: Principal Investigator, John E. Lewis, Associate Professor of Psychiatry and Behavioral Sciences, University of Miami
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20110168
Record Dates: First submitted 2012-05-09; First posted 2012-05-11 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Depression
Keywords: mild moderate treatment-resistant depression; magnesium sulfate
MeSH Terms: conditions — Depression | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magnesium sulfate crossover (Experimental): IV infusion of magnesium sulfate followed by 5-day washout period and crossover to 5% dextrose (placebo)
  Interventions: Dietary Supplement: Magnesium sulfate
- Placebo crossover (Placebo Comparator): IV infusion of 5% dextrose with 5 day washout and crossover to magnesium sulfate
  Interventions: Dietary Supplement: Magnesium sulfate

INTERVENTIONS:
Dietary Supplement: Magnesium sulfate — 4 grams magnesium sulfate in 100 ml IV over 4 hours

SUMMARY:
The proposed study is a 1-week, randomized, double-blind, placebo-controlled, trial to evaluate the efficacy of an IV infusion of magnesium sulfate on symptoms of treatment resistant mild and moderate depression in 20 males and females (21-70 years of age). Participants will be assessed at screening/baseline, day 1, day 2, day 7, and day 8. Each subject will be randomized in a double-blind fashion to receive either IV infusion of magnesium sulfate or 5% dextrose followed by a washout period of 5 days then crossover to receive either IV infusion of 5% dextrose or magnesium sulfate.

DETAILED DESCRIPTION:
Purpose:

1. To determine the magnesium deficient status in treatment-resistant mild and moderate depression patients via 24-hour urine magnesium assessment before and after IV magnesium infusion.
2. Correlation of intracellular magnesium (EXATEST), urine magnesium, and serum magnesium as well as sensitivity to the IV magnesium infusion.
3. To assess the effectiveness of magnesium sulfate infusion on treatment resistant mild and moderate depression patients.

Objectives:

Primary:

1. To investigate the magnesium deficient status in treatment-resistant mild and moderate depression patients via assay of 24-hour urine magnesium, blood magnesium, and EXATEST of intracellular magnesium of epithelial cells before and after IV infusion.
2. To assess the effectiveness of the magnesium sulfate infusion on the mean change in scores on the Hamilton Rating Scale for Depression and the Patient Health Questionnaire (PHQ-9) for depression.

Secondary:

1. To correlate the levels of magnesium with the scores on the Hamilton Rating Scale for Depression and the Patient Health Questionnaire (PHQ-9) for depression.

ELIGIBILITY:
Inclusion Criteria:

1. Potential participants must be English speaking.
2. Between the ages of 21 and 70.
3. Overall healthy and have no difficulty with digestion or absorption of food
4. Have treatment-resistant depression defined as failure of clinical improvement after 6 weeks with an approved dose of a Selective Serotonin Uptake Inhibitor (SSRI), Serotonin-Norepinephrine Reuptake Inhibitor (SNRI), Selective Noradrenaline Reuptake Inhibitor (NRI), tricyclic antidepressant, or bupropion.
5. Willing to provide informed consent to participate in the study.
6. Willing and able to comply with all study procedures and data recording obligations for the entire length of the study.
7. Able and willing to abstain from alcohol from 48 hours prior to the first intravenous infusion until after completion of the post-treatment follow-up visit (Day 2) and from 48 hours prior to the second intravenous infusion until after completion of the post-treatment follow-up visit (Day 8).
8. If currently taking an SSRI for more than 90 days, have maintained the same dose for the past 90 days.
9. A non-smoker or have quit smoking at least 6 months ago.

Exclusion Criteria:

1. Currently enrolled (or have been in the last 30 days) in another research trial for investigative nutritional or other therapies thought to have an impact on depression.
2. Currently taking a medication or nutritional supplement containing more than 100% RDA of magnesium (for women over age 31, it is 320 mg/day and for men over age 31, it is 420 mg/day) and unable to discontinue using it 14 days prior to the Day 1 visit. (Current use must be stopped 2 weeks before enrolling in the study and during trial.)
3. Diagnosed with any medical condition, including diabetes, cardiovascular disease, pulmonary, renal, endocrine, hepatic, neurologic, psychiatric (except for depression), immunologic, hematologic, gastrointestinal, or metabolic disease requiring medical treatment that would preclude participation in the study.
4. Taking Digoxin (used to treat congestive heart failure and to slow the heart rate in patients with atrial fibrillation.
5. Taking penicillamine (also known as Cuprimine or Depen for Wilson's disease or rheumatoid arthritis).
6. Taking any antibiotic (including tetracycline or a quinolone).
7. Taking any psychotropic medication for any indication, except sedatives for sleep such as Zolpidem, in addition to the SSRI, SNRI, NRI, tricyclic antidepressant, or bupropion in the course of treatment for your depression.
8. Taking a SSRI, SNRI, NRI, tricyclic antidepressant, or bupropion for less than 90 days or unable to maintain the same therapeutic regimen throughout the study duration.
9. A history of any medical or surgical procedure that would preclude participation in the study.
10. Diagnosed with gastrointestinal disorders that could lead to uncertain resorption of the study supplements.
11. Pregnant, plan to become pregnant, or currently breast feeding.
12. Unwilling to avoid pregnancy (use medically-acceptable birth control method during the study with at least one method for the period of one month prior to beginning of the study until at least three months after study completion or are surgically sterile or postmenopausal (at least 12 months without a period).
13. Systolic blood pressure >160 mmHg or diastolic blood pressure >90 mmHg.
14. Had any of the following abnormal laboratory test values: (a) bilirubin > 2x upper normal limit, (b) AST and ALT > 2x upper normal limit, (c) serum creatinine > 1.5 mg/dl, (d) blood glucose below 80 mg/dl or above 110 mg/dl, (e) calcium level < 8.6 mg/dl, or (f) triglycerides >200 mg/dl.
15. Currently undergoing any chemotherapy or radiation treatment for cancer, have an active malignancy, or have had within the past 5 years any type of malignancy, other than non-melanomatous skin malignancies.
16. A history of substance abuse (e.g., alcohol, opiates, benzodiazepines, or amphetamines).
17. Currently consume more than 6 standard alcoholic drinks a week (A standard alcoholic drink is defined as one bottle/can of beer, one glass of wine, or one ounce of hard liquor.).
18. Diagnosed with a terminal illness.
19. Donated blood in the last 30 days.
20. Any severe, acute illness within the last five days.
21. Have a pacemaker or internal medical device.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Magnesium levels in treatment resistant mild and moderate depression | 8 days
  To investigate the magnesium deficient status in treatment-resistant mild and moderate depression patients via assay of 24-hour urine magnesium, blood magnesium, and EXATEST of intracellular magnesium of epithelial cells before and after IV infusion.
Self reported depression measures | 8 days
  To assess the effectiveness of the magnesium sulfate infusion on the mean change in scores on the Hamilton Rating Scale for Depression and the Patient Health Questionnaire (PHQ-9) for depression.

SECONDARY OUTCOMES:
Correlation of magnesium levels with self reported measures of depression | 8 days
  To correlate the levels of magnesium with the scores on the Hamilton Rating Scale for Depression and the Patient Health Questionnaire (PHQ-9) for depression

CONTACTS AND LOCATIONS:
Overall Officials: John Lewis, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Clinical Research Building, Miami, Florida, United States